CLINICAL TRIAL: NCT00883597
Title: Sidestream Dark-Field Imaging of the Intestinal Microcirculation in Clinical Sepsis: The Impact of Activated Protein C Therapy
Brief Title: Sidestream Dark-Field (SDF) Imaging of the Intestinal Microcirculation
Status: Completed | Type: Observational
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Nova Scotia Health Research Foundation (Other Government)
Responsible Party: Sponsor
Other Study IDs: CDHA-RS/2009-311
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Controls: Patients with ileostomy.
- Standard Sepsis Treatment: Patients with ileostomy and sepsis

SUMMARY:
Sepsis is the most frequent cause of death in critically ill patients in non-coronary care Intensive Care Units in the developed world. Microcirculatory disturbances are central to the development of the disorder, leading to organ dysfunction, multi-organ failure and fatal outcome.

In particular the intestinal microcirculation is impaired early in the course of the disease. This may result in a breakdown of the gut barrier function with translocation of bacteria and their toxins into the systemic circulation, thus sustaining a "gut derived" septic state. Therefore, the impaired intestinal microcirculation has been suggested to act as the "motor of multiple organ failure" in sepsis.

The aim of the project is to evaluate a new diagnostic tool and the impact of Activated Protein C administration on the intestinal microcirculation in patients with severe sepsis and compare the findings with septic patients who are not candidates for APC therapy and healthy patients post bowel surgery using an innovative diagnostic tool (side stream dark-field imaging, SDF).

ELIGIBILITY:
Inclusion Criteria:

* ileostomy, no infection at the site of stoma, informed consent.
* diagnosed sepsis according to American College of Chest Physicians/Society of Critical Care Medicine criteria13.
* indication for treatment according to hospital guidelines

Exclusion Criteria:

* infection at the site of stoma,
* moribund patients

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to ICU with sepsis and ileostomy
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Microvascular Flow Index (MFI) | 6 hours after treatment

SECONDARY OUTCOMES:
Leukocyte - endothelial cell interactions, red blood cell velocity | 6 hours after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Elizabeth II Health Sciences Cetnre, Halifax, Nova Scotia, Canada